

| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | | |
|---|---|---|---|
| Туре | Version | Document Identifier | Effective Date |
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 | |
| Reason For Issue | | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018



# STATISTICAL REPORTING AND ANALYSIS PLAN

A RANDOMIZED, EXAMINER BLIND, CROSSOVER, IN SITU EROSION STUDY TO INVESTIGATE THE EFFICACY OF AN EXPERIMENTAL DENTIFRICE IN REMINERALIZATION OF PREVIOUSLY SOFTENED ENAMEL COMPARED TO PLACEBO DENTIFRICE

Protocol Number: 208166

Phase: 3

Property of GSK Consumer Healthcare
Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of GSK
Template Version Effective: 15-Jul-2017




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

# **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Amendment 1 | 27-Feb-2018 | Blinded data review of surface micro hardness data helped to identify a discrepancy between clinical protocol and analytical protocol. Following that identification, an administrative letter (#3-22FEB2018) was issued to correct that discrepancy. Therefore, 208166 Statistical Report and Analysis Plan is amended to reflect this administrative change. The following text from section 4.4.1.2 will be amended: Old text: The baseline surface micro hardness and first demineralization level (E1) will not be included in the model as covariates as the samples will be preselected so that each sample has a measurement of 43 +/-3 µm (at baseline, B) and 120 ± 20 µm (after the first erosive challenge, E1). New text: The baseline surface micro hardness and first demineralization level will not be included in the model as covariates as the samples will be preselected so that each sample has a measurement of 43 +/-3 µm at baseline (B) and 10-20 µm greater than the baseline after the first erosive challenge (E1). |
| Analysis Plan | 20-Dec-2017 | Not applicable (N/A) |

Amendments incorporate all revisions to date.

GlaxoSmithKline Consumer Healthcare 



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

| Ta | | f contents | | |
|---|---|---|---|---|
| | | _ | Ÿ | |
| | | - | | |
| 1 | Sum | - | Protocol Information | |
| | 1.1 | • | ign | |
| | 1.2 | Study Obj | ectives | 7 |
| | 1.3 | Treatment | S | 8 |
| | 1.4 | Sample Siz | ze Calculation | 9 |
| 2 | Planr | ed Analyses | | 9 |
| | 2.1 | Interim Ar | nalysis | 9 |
| | 2.2 | Final Anal | yses | 10 |
| 3 | Cons | iderations for | r data analyses and Data Handling Conventions | 10 |
| | 3.1 | Baseline D | Definition | 10 |
| | 3.2 | Subgroups | /Stratifications | 10 |
| | 3.3 | Centers Po | ools | 10 |
| | 3.4 | Timepoint | s and Visit Windows | 10 |
| 4 | Data | Analysis | | 10 |
| | 4.1 | Population | s for Analysis | 11 |
| | | 4.1.1 | Subject Disposition | 11 |
| | | 4.1.2 | Protocol Deviations | 11 |
| | | 4.1.3 | Analysis Populations | 12 |
| | 4.2 | Subject De | emographics and Other Baseline Characteristics | 13 |
| | | 4.2.1 | Demographic Characteristics | 13 |
| | | 4.2.2 | General Medical History | 13 |
| | 4.3 | | s (Study Drug, Rescue Medication, other Concomitant Therapies, ee) | 13 |
| | | 4.3.1 | Study Product Compliance and Exposure | 13 |
| | | 4.3.2 | Prior and Concomitant Medication | 13 |
| | 4.4 | Analysis o | f Efficacy | 14 |
| | | | Primary Efficacy Endpoint | |
| | | | Secondary Efficacy Variables | |
| | | | Handling of Missing Values/Censoring/Discontinuations | |
| | 4.5 | | f Secondary Objectives | |
| | | - | - · | |

GlaxoSmithKline Consumer Healthcare 



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

| | | 4.5.2 | Exploratory Efficacy Variables | 17 |
|-----|------|------------|----------------------------------------------|----|
| | 4.6 | Analys | is of Safety | 18 |
| | | 4.6.1 | Adverse Events and Serious Adverse Events | 18 |
| | | 4.6.2 | Other Safety Variables | 19 |
| | 4.7 | Analys | is of Other Variables | 20 |
| 5 | Chan | ges to the | e Protocol Defined Statistical Analysis Plan | 20 |
| | Appe | endix 1: S | Subgroups | 21 |
| | | | Center pools in multicenter studies | |
| | Appe | endix 3: N | Major Protocol Deviations | 21 |
| Att | | | of Data Display | |
| | | | emplates for Tables, Figures & Listings | |



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

**Glossary** 

| Glossary | |
|----------|----------------------------------------------|
| AE | adverse event |
| ARR | acid resistance ratio |
| ANOVA | analysis of variance |
| BDRM | blind data review meeting |
| CI | confidence interval |
| EFU | Enamel fluoride uptake |
| GSKCH | GlaxoSmithKline Consumer Healthcare |
| IRB | institutional review board |
| ITT | intent-to-treat |
| MedDRA | medical dictionary for regulatory activities |
| OHT | oral hard tissue |
| OST | oral soft tissue |
| PDMP | Protocol Deviation Management Plan |
| PP | per protocol |
| RER | relative erosion resistance |
| RLR | review listing requirement |
| SD | standard deviation |
| SE | standard error |
| SMHR | surface micro hardness recovery |
| SOC | System Organ Class |
| TEAE | treatment emergent adverse event |
| TLF | tables, listings and figures |



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

The purpose of this Statistical Reporting and Analysis Plan is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 208166.

## 1 Summary of Key Protocol Information

The aim of this study is to investigate the performance of an experimental dentifrice formulation in promoting enamel remineralization and inhibiting post-treatment enamel demineralization in an *in situ* erosion model, in comparison with a fluoride-free placebo and with a marketed competitor dentifrice product.

## 1.1 Study Design

This will be a randomized, controlled, single center, single- blind (to the dental examiner and specimen analysts), 3 period, 3 treatment, cross-over, *in situ* design which consists of placing pre-eroded bovine enamel specimens intra orally using a palatal appliance and testing the remineralizing performance of the experimental, comparator and placebo dentifrices 2 and 4 hours post treatment application, based on surface micro hardness measurements. This study will be carried out in healthy adults with a maxillary dental arch suitable for the retention of the palatal appliance.

There will be 4 visits, 1 screening visit to assess subject eligibility and 3 treatment visits to assess product efficacy, where the treatment product will be dispensed and used under the supervision of a suitably trained study site personnel. Prior to each treatment visit, there will be a washout period of a minimum of 3 days. During this period subjects will use their own dentifrice for at least one day, and a fluoride free dentifrice (provided) for two days prior to the next scheduled visit (including in the morning of the scheduled visit) to minimize any carry-over effects of the fluoride toothpaste.

The overall study design sequence of events is sketched in the figure below:



GlaxoSmithKline Consumer Healthcare Confidential




| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

# 1.2 Study Objectives

| Objectives | Endpoints |
|---|---|
| Primary Objective | |
| To investigate the efficacy of an | %SMHR after 4 hours intraoral phase |
| experimental dentifrice containing 1150 | following a single exposure. |
| ppm fluoride and 5% KNO <sub>3</sub> to enhance | |
| remineralization of enamel relative to a | |
| fluoride free placebo dentifrice. | |
| Secondary Objectives | |
| Efficacy | |
| To investigate the efficacy of an | %RER after 4 hours intraoral phase |
| experimental dentifrice containing 1150 | following a single exposure. |
| ppm fluoride and 5% KNO <sub>3</sub> to inhibit | |
| demineralization of enamel relative to a | |
| fluoride free placebo dentifrice. | |
| To investigate the efficacy of an | EFU after 4 hours intraoral phase following a |
| experimental dentifrice containing 1150 | a single exposure. |
| ppm fluoride and 5% KNO <sub>3</sub> to promote | |
| fluoride uptake in ename relative to a | |
| fluoride free placebo dentifrice. | |
| To investigate the efficacy of an | %SMHR, %RER and EFU after 4 hours |
| experimental dentifrice containing 1150 | intraoral phase following a single exposure. |
| ppm fluoride and 5% KNO <sub>3</sub> to enhance | |
| remineralization, to inhibit | |
| demineralization and to promote fluoride | |
| uptake in enamel relative to a benchmark | |
| comparator containing 1100 ppm fluoride | |
| (Crest Pro Health). | |
| Safety | |
| To evaluate the oral tolerance of an | Proportion of treatment emergent oral |
| experimental dentifrice containing 1150 | adverse events post 4 hours intraoral |
| ppm fluoride and 5% KNO <sub>3</sub> following a | exposure. |
| single brushing event. | |
| Exploratory Objectives | Exploratory Endpoints |
| To make all paired comparisons of the | %SMHR, %RER and EFU after 2 hours |
| efficacy of an experimental dentifrice | intraoral phase following a single exposure. |
| containing 1150 ppm fluoride and 5% | |
| KNO <sub>3</sub> after 2 hours of intraoral exposure | |
| to enhance remineralization of enamel, to | |
| inhibit demineralization of enamel and to | |

GlaxoSmithKline Consumer Healthcare 



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

| Objectives | Endpoints |
|---|---|
| promote fluoride uptake in enamel. | |
| To characterize the efficacy of the | Summary statistic table of ARR after 2 and 4 |
| experimental dentifrice containing 1150 | hours intraoral phase. |
| ppm fluoride and 5% KNO <sub>3</sub> ; the fluoride | |
| free placebo; and the benchmark | |
| comparator containing 1100 ppm (Crest | |
| Pro Health) after 2 and 4 hours of | |
| intraoral exposure on resistance to acid | |
| challenge. | |

**Abbreviations:** SMHR: Surface micro hardness recovery, RER: Relative erosion resistance, EFU: Enamel fluoride uptake, ARR: Acid resistance ratio

#### 1.3 Treatments

This is a single blind study, with the examiner and specimen analyst being blind to the treatment each subject received. Given that it is almost impossible to ensure identical appearance, taste and packaging for the dentifrices evaluated in this study, the level of blindness for this study is described as 'examiner blind' only. All study products (experimental, comparator and placebo dentifrices) will be over-wrapped in white vinyl to maintain the study blind as much as possible.

Subjects will be assigned to study product sequence in accordance with the randomization schedule generated by Inventiv Health under the supervision of the Biostatistics Department, GlaxoSmithKline Consumer Health (GSK CH), prior to the start of the study, using a validated program. Subjects will be randomized in a Williams square design balanced for first period carryover.

The details of the study treatments is outlined in below table

| | Test Product | Comparator<br>Product | Placebo Product |
|---|---|---|---|
| Product Name | Experimental dentifrice containing | Crest ProHealth<br>Sensitivity & | Fluoride free placebo containing 5% KNO <sub>3</sub> |
| | 0.254% w/w sodium<br>fluoride (1150 ppm<br>fluoride) and 5% | Enamel Shield<br>containing 0.454%<br>w/w stannous | (0 ppm fluoride); plus<br>0.25% PVM/MA<br>copolymer and 2.5% |
| | KNO <sub>3</sub> ; plus 0.25%<br>PVM/MA<br>copolymer and 2.5%<br>sodium lactate | fluoride (1100 ppm<br>fluoride) | lactate |

GlaxoSmithKline Consumer Healthcare 



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

| Product<br>Formulation<br>Code (MFC) | CCI | Commercially<br>available (US<br>marketed) | CCI |
|---|---|---|---|
| Dose | 1.5 g | 1.5 g | 1.5 g |
| Route of<br>Administration | Oral | Oral | Oral |
| Dosing<br>Instructions | Subjects will apply a full ribbon of the allocated product and brush the buccal surfaces of their natural teeth for 25 timed seconds and then swish the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the subjects will gently rinse their mouths with 15 mL of tap water for 10 seconds before expectorating again | | |

# 1.4 Sample Size Calculation

A sufficient number of healthy subjects will be screened so that up to 66 subjects are randomized to participate in the study to ensure 60 evaluable subjects complete the entire study.

A sample size of 60 subjects will be large enough to also detect a difference of 7.4 in RER with 80% power.

A sufficient number of healthy adult subjects will be selected from the Oral Health Research Institue's IRB approved database of previous research studies or from persons expressing interest in participating in research, and screened for participation.

# 2 Planned Analyses

# 2.1 Interim Analysis

No interim analysis is planned.

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

## 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and database has been locked.
- 3. All criteria for unblinding the randomization codes have been met and the randomization codes have been distributed.

# 3 Considerations for data analyses and Data Handling Conventions

#### 3.1 Baseline Definition

For Efficacy analyses:

Subject level baseline is defined as the latest assessment with a non-missing value before the first erosive challenge.

Period level baseline is defined as the latest assessment with a non-missing value the first erosive challenge for a given period.

Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 3.2 Subgroups/Stratifications

No stratification or subgrouping is planned for this study.

#### 3.3 Centers Pools

This is single centre study, therefore pooling of centers is not applicable.

## 3.4 Timepoints and Visit Windows

The study schedule should be followed as per protocol. Deviations from the study schedule with respect to visit timings and the amount of time the appliance was worn at each visit will be reviewed and significant deviations in timings classified as protocol deviations potentially affecting efficacy assessment. A time window non-compliance listing will be produced for blinded data review.

## 4 Data Analysis

Data analysis will be performed by inVentiv Health Clinical. The statistical analysis software used will be SAS version 9.4 (Studio) or higher.

GlaxoSmithKline Consumer Healthcare 



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Prior to database closure a blind data review meeting (BDRM) will be conducted in which various aspects of the trial will be discussed and agreed.

Unless otherwise described, all listings will be produced for all randomized subjects.

## 4.1 Populations for Analysis

#### 4.1.1 Subject Disposition

Screen failures are defined as subjects who consent to participate in the study but are never subsequently randomized. A summary of the number of subjects screened and the number of screen failures will be provided. Percentage calculation for screen failures will based on all screened subjects.

Subject disposition will be summarized as the number and percentage of subjects who complete the study, with the number who discontinue, broken down by reason for discontinuation. The percentages are based on the total number of subjects randomized. The table will also summarise the number and percent of subjects assigned to each analysis population (defined in Section 4.1.3). The summary will be presented by treatment group and overall (Table 14.1.1). In addition summary will be presented by sequence group, period and overall (Table 14.1.2).

Subject disposition including the subject status (completer, Yes/No), critical demographic data (age, sex and race) will be listed for randomized subjects (Listing 16.2.1.1) and non-randomized subjects (Listing 16.2.1.2) separately.

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. All deviations will be reviewed prior to unblinding and closure of the database to ensure all important deviations are captured and categorised.

The following will be taken into consideration when determing the protocol deviations with the potential to affect primay efficacy assessment.

- Deviation from the inclusion/exclusion criteria
- Use of prohibited medication before or during the study which is deemed to affect the assessment of efficacy.
- Significant non-compliance of product use.
- Significant non-compliance with the study schedule e.g., with regards to durations that appliances are worn.
- Significant deviation from planned time of an evaluation.
- Treatment not received in defined order.
- Any other reason identified which may affect the assessment of efficacy.

GlaxoSmithKline Consumer Healthcare Confidential




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Major deviations deemed to affect primary efficacy will be identified between the Biostatistician and Clinical Research Director or designee, before breaking the study blind and will be documented in the Population Definition Document. These will be excluded from the Per-Protocol (PP) analysis.

Minor deviations will be identified as those not classified as major deviations.

More details on protocol deviations can be found in the Protocol Deviation Management Plan (PDMP) of this study.

The number and percentage of subjects with any major protocol deviations and with each type of major protocol deviations will be presented by treatment (Table 14.1.3) and listed (Listing 16.2.2.1). Any minor protocol deviations will be listed similarly (Listing 16.2.2.2).

#### 4.1.3 Analysis Populations

Following analysis populations are defined.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened | All subjects who are screened | Disposition |
| Subjects | | |
| Randomized | All subjects who are randomized and may or | Protocol deviations |
| | may not receive the study treatment. | |
| Safety | Safety population includes all subjects who | Safety analysis |
| | are randomized and receive at least one dose | |
| | of study treatment during the study. Safety | |
| | population summaries will be presented by | |
| | treatment received. | |
| Intent-to-Treat | The primary population for efficacy | Efficacy analysis |
| (ITT) | assessment will be the (ITT) population, | |
| | defined as all subjects who are randomized, | |
| | receive the study treatment at least once and | |
| | provide at least one post-baseline (post | |
| | treatment) assessment of primary efficacy. | |
| | All ITT population summaries and analyses | |
| | will be presented by treatment randomized. | |
| PP | The PP population is defined as all subjects | Primary efficacy |
| | in the ITT population who have at least one | analysis |
| | assessment of the primary endpoint efficacy | (%SMHR) only |
| | considered unaffected by protocol violations. | |

Efficacy analysis on PP population will be performed only if there is more than 10% difference in the overall number of subjects between PP and ITT populations.

A decision on whether a PP analysis will be performed will be made prior to study unblinding. Subjects excluded from any of the analysis populations will be listed (Listing 16.2.3.1).

GlaxoSmithKline Consumer Healthcare 



| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

## 4.2 Subject Demographics and Other Baseline Characteristics

#### 4.2.1 Demographic Characteristics

Demographic and baseline characteristics summaries will be produced for the Safety Population (Table 14.1.4.1). ITT Population (Table 14.1.4.2), and PP Population (Table 14.1.4.3) (if PP analysis is performed).

Categorical demographic variables include sex, ethnicity and race, will be summarized by the number and percentage of subjects in each treatment group. The continuous demographic variable age (in years) and will be summarized by the mean, standard deviation (SD), median, minimum and maximum values. All summaries will be presented by overall.

All demographic information will be listed for randomized subjects (Listing 16.2.4.1).

#### 4.2.2 General Medical History

Medical history and current medical conditions for all randomized subjects will be listed (Listing 16.2.4.2) with start date and end date or ongoing at the first application of study drug.

# 4.3 Treatments (Study Drug, Rescue Medication, other Concomitant Therapies, Compliance)

Treatment compliance will also be listed for the blinded data review and specified in the review listing requirement (RLR) document.

#### 4.3.1 Study Product Compliance and Exposure

Subjects will complete diary cards during the 2 days of washout period prior to the treatment visit. Study product compliance will be listed (Listing 16.2.5.3).

#### 4.3.2 Prior and Concomitant Medication

Prior medications are defined as those stopped before the first administration of study drug. Any medication that has started prior to first dose of study drug and is still continuing is termed as concomitant medication.

Concomitant medication is also defined as any medication taken between the date of first dose of study drug and the date of last dose of study drug.

In this crossover trial, medications will be assigned to the treatment group based on the treatment being received at that date. Medications with a date time between treatments periods will be assigned to the treatment received in the previous period. Medications with a date after last treatment or the end of the study will be assigned to the treatment taken in the last period.

There will be no imputation of unknown dates. However if the start date is unknown, then it will be assumed to concomitant (all treatment periods) unless the partial start date or stop date indicates differently.

GlaxoSmithKline Consumer Healthcare Confidential




| <b>Document Name</b> | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Prior and concomitant medications and siginificant non-drug therapies will be listed by subject, with preferred term, indication, dose, dose form, frequency, route, start date, end date or ongoing and start day relative to first dose of study drug (Listing 16.2.5.1 and Listing 16.2.5.2).

## 4.4 Analysis of Efficacy

#### 4.4.1 Primary Efficacy Endpoint

#### 4.4.1.1 Primary Efficacy Endpoint Definition

The primary efficacy endpoint is %SMHR after 4 hours of remineralization.

Definition of primary variable: % SMH recovery = [(E1-R)/(E1-B)] \* 100

 $B = indentation length (\mu m)$  of sound enamel at baseline

 $E1 = indentation length (\mu m)$  after first erosive challenge

 $R = indentation length (\mu m)$  after in situ remineralization

Per subject %SMHR will be determined from the %SMHR calculated for each specimen using five indentations measurements per specimen, averaged across the four specimens at 4 hours. Therefore, a single observation per treatment for each subject will be used in the statistical analyses. If a subject is missing an enamel specimen, the mean will be computed over the available enamel specimens.

#### 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

The primary comparison of this study is the 1150 ppm fluoride experimental dentifrice versus the fluoride free placebo (0 ppmF) in %SMHR at 4 hours and must be statistically significant to meet the success criteria.

The extent of remineralization will be calculated as the % recovery in SMH (%SMHR), which is calculated from the enamel indentation length at baseline, after the first erosive challenge and after the *in situ* remineralization phase after 4 hrs of intraoral phase.

Statistical testing of all endpoints in this study will be conducted at a two-sided significance level of 0.05. As a primary objective has been defined prior to analysis, there will be no adjustment for multiple comparisons. The null and alternative hypotheses are

- H<sub>0</sub>: there is no difference between treatment groups;
- H<sub>1</sub>: there is a difference between treatment groups.

GlaxoSmithKline Consumer Healthcare Confidential




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

The analysis of variance (ANOVA) will be used to analyze the treatment difference. The ANOVA model will include fixed factors for study period and treatment, and a random effect for subject. The baseline SMH and first demineralization level will not be included in the model as covariates as the samples will be preselected so that each sample has a measurement of  $43 + 1/-3 \mu m$  at baseline (B) and  $10-20 \mu m$  greater than the baseline after the first erosive challenge (E1).

Summary statistics including mean, standard deviation (SD), standard error (SE), median, min, max will be provided on the analysis population used for statistical analysis (Table 14.2.1.1) by treatment group.

Adjusted means of two treatments and treatment difference will be provided together with 95% confidence interval (CI) and p-values (Table 14.2.1.1) by treatment group.

The assumption of residual normality and variance homogeneity in ANOVA analysis will be investigated through residual plots. If violated, a nonparametric method (paired Wilcoxon Sign Rank test) will be performed. If the violation is caused by extreme values, a sensitivity analysis will be conducted by removing the extreme values and same analysis will be repeated without those extreme values. If nonparametric test is performed and the inferences on treatment comparisons are similar to that of ANOVA, both sets of results will be reported and the emphasis will be made on the ANOVA results. Otherwise, nonparametric results will be used to draw conclusions.

A Bar Chart (Figure 14.2.1.5) with Error Bars (±SD) will be created.

#### 4.4.1.3 Supportive Analyses

If there are more than 10% differences in the overall number of subjects between PP and ITT populations, a PP analysis will be performed for primary efficacy variable. This analysis would be considered as supportive analysis (Table 14.2.1.3).

A summary table (Table 14.2.1.4) for derived specimens by timepoint and treatment groups will be provided.

#### 4.4.2 Secondary Efficacy Variables

Secondary efficacy variables of the study are defined in section 4.5.

#### 4.4.3 Handling of Missing Values/Censoring/Discontinuations

Missing data will not be replaced or imputed. Dropouts will be included in analyses up to the point of discontinuation.

#### 4.5 Analysis of Secondary Objectives

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

The treatment difference, SE and 95% CI will be presented for all of the comparisons however the p-values for these secondary comparisons will only be presented if the primary comparison is statistically significant.

Same model and analysis methods of primary efficacy endpoint will be conducted for all secondary efficacy endpoints.

#### 4.5.1.1 Percent Relative Erosion Resistance (RER) after 4 Hours

The %RER is calculated based on the indentation length at baseline, after the first and the second erosive challenge after 4 hours.

% Relative Erosion Resistance = [(E1-E2)/(E1-B)] \* 100

B= Indentation length (μm) of sound enamel at baseline

E1= Indentation length (μm) after first erosive challenge

E2= Indentation length (µm) after second erosive challenge

Per subject % RER will be determined from the % RER calculated for each specimen using five indentations measurements per specimen, averaged across the four specimens at 4 hours. Therefore, a single observation per treatment for each subject will be used in the statistical analyses. If a subject is missing an enamel specimen, the mean will be computed over the available enamel specimens.

Summary statistics including mean, SD, SE, median, min, max will be provided on the analysis population used for statistical analysis (Table 14.2.2.1) by treatment group. Adjusted means of two treatments and treatment difference will be provided together with 95% confidence interval (CI) and p-values (Table 14.2.2.1) by treatment group. As a primary objective has been defined prior to analysis, there will be no adjustment for multiple comparisons.

A Bar Chart (Figure 14.2.2.3) with Error Bars (±SD) will be created.

#### 4.5.1.2 Enamuel Fluoride Uptake (EFU) after 4 Hours

EFU is assessed by the microdrill enamel biopsy, and is determined after 4 hours *in situ* remineralization period but before the second extra-oral erosive challenge. This measurement will provide with micrograms of fluoride per square centimeter (μg F/cm²).

Per subject EFU score will be calculated as follows: microdrill samples from each enamel specimen will be pooled and a value for fluoride content per enamel specimen determined. These values will be averaged across the four enamel specimens for each subject and time point to produce the subject-wise mean enamel fluoride uptake.

Summary statistics including mean, standard deviation (SD), standard error (SE), median, min, max will be provided on the analysis population used for statistical analysis (Table 14.2.3.1) by treatment group. Adjusted means of two treatments and treatment difference will

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

be provided together with 95% CI and p-values (Table 14.2.3.1) by treatment group. As a primary objective has been defined prior to analysis, there will be no adjustment for multiple comparisons.

A Bar Chart (Figure 14.2.3.3) with Error Bars (±SD) will be created.

#### 4.5.2 Exploratory Efficacy Variables

Exploratory variables of the study are listed below. Unless not stated otherwise same model and analysis methods will be conducted as for the secondary endpoints.

#### 4.5.2.1 Percent Surface Microhardness Recovery after 2 Hours

The extent of remineralization will be calculated as the % recovery in SMH, which is calculated from the enamel indentation length at baseline, after the first erosive challenge and after the *in situ* remineralization phase after 2 hours of intraoral phase.

Summary statistics including mean, SD, SE, median, min, max will be provided on the analysis population used for statistical analysis (Table 14.2.1.2) by treatment group. Adjusted means of two treatments and treatment difference will be provided together with 95% CI and p-values (Table 14.2.1.2) by treatment group. As a primary objective has been defined prior to analysis, there will be no adjustment for multiple comparisons.

A Bar Chart (Figure 14.2.1.5) with Error Bars ( $\pm$ SD) will be created.

#### 4.5.2.2 Percent Relative Erosion Resistance after 2 Hours

This end point aims to test whether the formulations prevents enamel demineralization after the 2 hours intra oral remineralization phase as per a second erosion challenge. The %RER is calculated based on the indentation length at baseline, after the first and the second erosive challenge after 2 hours.

Summary statistics including mean, SD, SE, median, min, max will be provided on the analysis population used for statistical analysis (Table 14.2.2.2) by treatment group. Adjusted means of two treatments and treatment difference will be provided together with 95% CI and p-values (Table 14.2.2.2) by treatment group. As a primary objective has been defined prior to analysis, there will be no adjustment for multiple comparisons.

A Bar Chart (Figure 14.2.2.3) with Error Bars (±SD) will be created.

#### 4.5.2.3 Enamuel Fluoride Uptake (EFU) after 2 Hours

EFU is assessed by the microdrill enamel biopsy, and is determined after 2 hours *in situ* remineralization period but before the second extra-oral erosive challenge. This measurement will provide with micrograms of fluoride per square centimeter (μg F/cm<sup>2</sup>).

Summary statistics including mean, SD, SE, median, min, max will be provided on the analysis population used for statistical analysis (Table 14.2.3.2) by treatment group. Adjusted means of two treatments and treatment difference will be provided together with 95% CI and

GlaxoSmithKline Consumer Healthcare Confidential




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

p-values (Table 14.2.3.2) by treatment group. As a primary objective has been defined prior to analysis, there will be no adjustment for multiple comparisons.

A Bar Chart (Figure 14.2.3.3) with Error Bars (±SD) will be created.

#### 4.5.2.4 Acid Resistance Ratio (ARR)

The ARR measures acid resistance of the treated enamel after 2 and 4 hours intraoral phase. It is calculated based on the indentation length after the second erosive challenge and the *in situ* remineralization phase, and after the first erosive challenge and baseline.

The ARR will be calculated as follows: ARR = 1 - [(E2-R)/(E1-B)]

B= Indentation length (μm) of sound enamel at baseline

E1= Indentation length (μm) after first erosive challenge

E2= Indentation length (μm) after second erosive challenge

 $R = indentation length (\mu m)$  after in situ remineralization

Only summary statistics including mean, SD, SE, median, min, max will be provided by randomized treatment group (Table 14.2.4.1, Table 14.2.4.2) for 4 hours and 2 hours respectively.

A Bar Chart (Figure 14.2.4.3) with Error Bars ( $\pm$ SD) will be created.

## 4.6 Analysis of Safety

#### 4.6.1 Adverse Events and Serious Adverse Events

All summaries of safety will be performed using the safety population and will be analyzed based on treatment actually received. No formal statistical testing will be performed on summary comparisons related to safety related measurements.

All AEs will be coded using the medical dictionary for regulatory activities (MedDRA). AEs will be classified by system organ class (SOC) and by preferred term (PT). In addition, prior to database lock all AEs will be reviewed by the Clinical Research Director (or designee) and categorized as either oral or non-oral. Safety will be assessed based on any oral AEs (this includes those that are identified as treatment emergent oral soft tissue (OST) abnormalities and spontaneously reported oral AEs). Any new or worsening OST condition that occurs after the OST examinations at Screening will be recorded as an AE.

In this crossover trial, events will be assigned to the treatment group based on the treatment being received at the onset of the event. TEAEs with an onset date time between treatments perods will be assigned the treatment received in the previous period. TEAEs with an onset after last treatment or the end of the study will be assigned to the treatment taken in the last period. If an emergent AE continues to another treatment period and worsens, the AE will be

GlaxoSmithKline Consumer Healthcare Confidential




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

considered emergent in both the period in which it started and also the period in which it worsened.

AEs will be summarized using descriptive statistics (frequency tables) by treatment group. Summary tables will indicate both the number of events and the number (percent) of subjects involved. Summaries of AEs will also include TEAEs unless otherwise noted. TEAEs are defined as new AEs that occur on or after the date/time of the first supervised use of the randomized treatment (or events aggravated in severity following treatment). Events with an onset date/time prior to first use of a treatment will be considered as non-treatment emergent.

The following summary tables and listings will be presented by treatment group.

- Table of Treatment emergent AEs by SOC and PT (Table 14.3.1.1)
- Table of Treatment emergent AEs by Oral/Non-Oral and PT (Table 14.3.1.2)
- Table of treatment emergent treatment related AEs by SOC and Preferred Term (Table 14.3.1.3).
- Table of treatment emergent treatment related AEs by Oral/Non-Oral and Preferred Term (Table 14.3.1.4).
- Table of treatment emergent AEs by intensity and Preferred Term.
   (Table 14.3.1.5).
- Listing of all AEs (including all subjects: Listing 16.2.7.1 for all randomized subjects; Listing 16.2.7.2 for non-randomized subjects).
- Listing of death (Listing 14.3.2.1).
- Listing of serious AEs (Listing 14.3.2.2) (if there are more than 5 treatment emergent serious AEs (SAEs) a table (Table 14.3.1.6) will be produced instead by SOC and PT).
- Listing of treatment emergent AEs leading to withdrawal (Listing 14.3.2.3).
- Listing of treatment emergent AEs classified as oral (Listing 14.3.2.4).
- Listing of non-fatal serious treatment emergent AEs (Listing 14.3.2.5) (only produced if there are more than 5 SAEs).

In the event that there is nothing to report a null listing will be produced.

#### 4.6.2 Other Safety Variables

A listing (Listing 16.2.7.3) for incidents will be produced. A table (Table 14.4.1.1) for OST will be produced for changes in abnormality pre- and post treatment. In addition a listing (Listing 16.2.9.2) for oral hard tissue (OHT) and OST (Listing 16.2.9.1) will be displayed.

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

# 4.7 Analysis of Other Variables

Not applicable.

# 5 Changes to the Protocol Defined Statistical Analysis Plan

There are no changes to the protocol-planned statistical analyses.

## **Top-line Summary:**

For the top-line report selected outputs will be produced as documented in the attached worksheet excel file.




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Appendix 1: Subgroups

Not Applicable

Appendix 2: Center pools in multicenter studies

Not Applicable

# **Appendix 3: Major Protocol Deviations**

Protocol deviations will be tracked by the study team throughout the conduct of the study. More details on protocol deviations can be found in the Protocol Deviation Management Plan (PDMP) of this study.

All deviations will be reviewed prior to study unblinding and closure of the database. Details will be given in the populations' definitions document.

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

208166

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

# **Attachment 1: List of Data Display**





| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Sodium fluoride and potassium nitrate 208166 Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

# Appendix 4: Templates for Tables, Figures & Listings

The following provides detail of the treatment labels to be used on the table, figure and listings and and general footnotes. The treatment labels will be specified as follows:

Test Product Comparator Product Placebo Product

If there are no data to display generate a null table or listing.

Add following footnote to all TFLs:

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166 Program Run Date:xxxx
Table 14.1.1

Subject Disposition by Treatment Group Across Study Treatment Periods  ${\tt All \ Screened \ Subjects}$ 

All Screened Subjects (N=xxx)

| | Test Product | Comparator Product | Placebo Product | Overall |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| TOTAL SUBJECTS SCREENED | | | | xxx |
| SUBJECTS NOT RANDOMIZED | | | | xxx |
| DID NOT MEET STUDY CRITERIA | | | | xxx (xx,x) |
| ADVERSE EVENT | | | | xxx (xx.x) |
| LOST TO FOLLOW UP | | | | xxx (xx,x) |
| PROTOCOL VIOLATION | | | | xxx (xx.x) |
| WITHDRAWAL OF CONSENT | | | | xxx (xx,x) |
| OTHER | | | | xxx (xx.x) |
| UBJECTS RANDOMIZED | xxx | xxx | xxx | xxx |
| COMPLETED STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT COMPLETE STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ADVERSE EVENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| LOST TO FOLLOW-UP | xxx (xx,x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATION | xxx (xx,x) | xxx (xx,x) | xxx (xx,x) | xxx (xx,x) |
| WITHDRAWAL OF CONSENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| OTHER | xxx (xx.x) | xxx (xx.x) | (xxx) (xxx) | xxx (xx.x) |
| SAFETY POPULATION | | | | xxx (xx,x) |
| TT POPULATION | | | | xxx (xx.x) |
| P POPULATION | | | | xxx (xx.x) |

For categories under 'Subjects Not Randomized' percentages will be calculated using the number of 'All Screened Subjects' as the denominator. Percentages under the 'Subjects Randomized' categories will be computed using number of subjects randomized as the denominator.

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166

Program Run Date:xxxx

Table 14.1.2 Subject Disposition by Sequence Group and Period All Screened Subjects

All Screened Subjects (N=xxx)

| | | | Treatment Seque | ence | | | |
|---|---|---|---|---|---|---|---|
| | A/B/C | A/C/B | B/A/C | B/C/A | C/A/B | C/B/A | OVERALL |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| TOTAL SUBJECTS SCREENED | | | | | | | XX |
| SUBJECTS NOT RANDOMIZED: | | | | | | | XX |
| DID NOT MEET STUDY CRITERIA | | | | | | | XX |
| ETC. | | | | | | | |
| SUBJECTS RANDOMIZED | XX | xx | xx | xx | xx | xx | xx |
| PERIOD X: | | | | | | | |
| STARTED PERIOD: | XX | XX | XX | XX | XX | XX | XX |
| COMPLETED | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| DID NOT COMPLETE: | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| DID NOT MEET STUDY CRITERIA | XX (XX,X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ETC. | | • • | | • • | | | |
| SAFETY POPULATION | xx | xx | xx | xx | XX | XX | XX |
| ITT POPULATION | XX | XX | XX | XX | XX | XX | XX |
| PP POPULATION | XX | XX | XX | XX | XX | XX | XX |

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD Page x of y



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


# Table 14.1.3 Incidence of Major Protocol Deviations All Randomized Subjects

Randomized Population (N=xxx)

| | | A/B/C | | A/C/B | 1 | B/A/C | | B/C/A | | C/A/B | | C/B/A | 01 | erall |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | (%) | n ( | %) | n | (%) | 1 | n (%) | n | (%) | n | (%) | n | (%) |
| SUBJECTS WITH AT LEAST ONE MAJOR PROTOCOL VIOLATION | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |
| MAJOR PROTOCOL VIOLATIONS NOT LEADING TO EXCLUSION FROM PP | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |
| VIOLATION REASON 1 | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |
| MAJOR PROTOCOL VIOLATIONS<br>LEADING TO EXCLUSION FROM PP<br>All VISITS | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |
| VIOLATION REASON 1 | xxx | (xx.x) | xxx | (xx,x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx,x) | xxx | (xx.x) |
| WEEK Y | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |
| VIOLATION REASON 1 | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD

Page x of y



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

| Protocol No. 208166 | |
|-------------------------------------------|------------------------------|
| | Table 14.1.4.1 |
| | Demographics Characteristics |
| | Safety Population |
| Safety Population (N=xxx) | |
| outer, ropulation (n mm) | Overall |
| | N (%) |
| SEX n (%) | |
| Male | xx (xx.x) |
| Female | xx (xx.x) |
| | , |
| RACE n (%) | |
| African American/African Heritage | xx (xx.x) |
| American Indian or Alaskan Native | xx (xx.x) |
| Asian - Central/South Asian Heritage | xx (xx.x) |
| Asian - East Asian Heritage | xx (xx.x) |
| Asian - Japanese Heritage | xx (xx.x) |
| Asian - South East Asian Heritage | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) |
| White - Arabic/North African Heritage | xx (xx.x) |
| White - White/Caucasian/European Heritage | xx (xx.x) |
| - | |
| ETHNICITY n (%) | |
| Hispanic or Latino | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) |
| AGE (YEARS) | |
| N | xx |
| MEAN | xx.x |
| SD | xx.xx |
| MEDIAN | xx.x |
| MINIMUM | xx |
| MAXIMUM | xx |

Page x of y

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Table 14.2.1.1

Statistical Analysis of Percent Surface Microhardness Recovery at 4 Hours by Treatment Group ITT Population

Intent-to-Treat Population (N=XX)

| | Test Product | Comparator Product | Placebo Product |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| n | xx | xx | xx |
| MEAN | x.xx | x.xx | x.xx |
| SD | x,xxx | x,xxx | x,xxx |
| SE | x,xxx | x,xxx | x,xxx |
| MEDIAN | x.xx | x.xx | x.xx |
| MINIMUM | X.xx | x.xx | x.xx |
| MAXIMUM | X.xx | x.xx | x.xx |
| ADJUSTED MEAN [1] | xx.xx | xx.xx | xx.xx |
| STANDAR ERROR | x.xxx | x.xx | x.xx |
| COMPARISON BETWEEN TREATMENTS | DIFFERENCE [1,2] | 95% CI [1] | P-VALUE [1] |
| TEST PRODUCT VS PLACEBO PRODUCT | x.xx | (xx.xx, xx.xx) | x.xxx |
| TEST PRODUCT VS COMPARATOR PRODUCT | x,xx | xx.xx, xx.xx) | x.xxxx |

<sup>[1]</sup> From ANOVA with fixed factors for study period and treatment, and a random effect for subject.

PPD Page x of y

<sup>[2]</sup> Difference is first-named treatment minus second-named treatment such that a positive difference favors the first named treatment.

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


 ${\tt Table~14.2.1.4}\\ {\tt Summary~Table~of~Indents~Measures~by~Timepoint~and~Treatment~Group}$ 

ITT Population

Intent-to-Treat Population (N=XX)

| | | | Indentation ler<br>sound enamel at 1 | | Indentation after firs | | | on length<br>nd Erosive | Indentation lengt | h after in situ |
|---|---|---|---|---|---|---|---|---|---|---|
| | | N | (B) (μm) | | Challenge | (E1) (μm) | Challenge | (E2) (μm) | Remineralizati | lon (R) (μm) |
| Timepoint | Treatment | | Mean | SE | Mean | SE | Mean | SE | Mean | SE |
| 4 Hours | Test Product | XX | xx.xx x, | xxx | xx.xx | x.xxx | xx.xx | x.xxx | xx,xx | x.xxx |
| | Comparator Product | XX | xx.xx x. | xxx | xx.xx | x.xxx | xx.xx | x.xxx | xx.xx | x.xx |
| | Placebo Product | XX | xx.xx x. | xxx | xx.xx | x.xxx | xx.xx | x.xxx | xx.xx | x.xxx |
| 2 Hours | Test Product | xx | xx.xx x. | xxx | xx.xx | x.xxx | xx.xx | x.xxx | xx.xx | x,xxx |
| | Comparator Product | XX | xx.xx x. | xxx | xx.xx | x.xxx | xx.xx | x.xxx | xx.xx | x.xxx |
| | Placebo Product | XX | xx.xx x. | xxx | xx.xx | x.xxx | xx.xx | x.xxx | xx.xx | x.xx |

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

Page x of v



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Sodium fluoride and potassium nitrate 208166 Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


 $\mbox{Figure 14.2.1.5} \\ \mbox{Bar Chart with Error Bars (+/- SD) for % Surface Microhardness Recovery} \\ \mbox{ITT Population}$ 



Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD Page v of v

Programming Note: Please adapt this figure with study specific informations and title specifications. Please include 2 hour and 4 hour in same figure.




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Intent-to-Treat Population (N=XX)

| | Test Product | Comparator Product | Placebo Product |
|---------|--------------|--------------------|-----------------|
| | (N=XX) | (N=XX) | (N=XX) |
| n | xx | xx | xx |
| MEAN | x.xx | x.xx | x.xx |
| SD | x,xxx | x,xxx | x,xxx |
| SE | x,xxx | x,xxx | x,xxx |
| MEDIAN | x,xx | x.xx | x.xx |
| MINIMUM | x.xx | x.xx | x.xx |
| MAXIMUM | x.xx | x.xx | x.xx |

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

Page x of y



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Sodium fluoride and potassium nitrate 208166 Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Table 14.3.1.1

Treatment Emergent Adverse Event by System Organ Class and Preferred Term Safety Population

| | Test | | Comparator Pr | oduct | Placebo | ) | | |
|---|---|---|---|---|---|---|---|---|
| SOC Preferred Term | Product (N=XX) | | (N=XX) | | Product (N=XX) | | Overall (N=XXX) | |
| _ | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT<br>LEAST ONE AE | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx,x) | xx | xx (xx.x) | xx |
| NUMBER OF SUBJECTS WITH NO AE | xx (xx,x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| SKIN AND SUBCUTANEOUS TISSUE | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| ERYTHEMA | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| DERMATITIS | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx,x) | xx | xx (xx.x) | xx |
| GASTROINTESTINAL SYSTEM | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| ABDOMINAL PAIN | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| DRY MOUTH | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| VOMITTING | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx,x) | xx | xx (xx.x) | xx |

Etc.

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

#### **PPD**

n (%) = Number (percent) of subjects nAE = Number of adverse events. SOC=System organ class



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166

Table 14.3.1.2

Treatment Emergent Adverse Event by Oral/Non-Oral and Preferred Term

Safety Population

Safety Population

Safety Population

| | Test Product (N=XX) | Comparator Product (N=XX) | Placebo Product (N=XX) | Overall (N=XXX) |
|---|---|---|---|---|
| Preferred Term | n (%) nAE | n (%) nAE | n (%) nAE | n (%) nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE TEAE | xx (xx.x) xx | xx ( xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| NUMBER OF SUBJECTS WITH NO TEAE | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| ORAL | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| SENSITIVITY OF TEETH | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ORAL MUCOSAL EXOLIATION | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx | xx (xx,x) xx |
| NON ORAL | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| BRONCHITIS | xx (xx.x) xx | xx (xx.x) xx | xx (xx,x) xx | xx (xx.x) xx |
| COUGH | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

n (%) = Number (percent) of subjects nAE = Number of adverse events.

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD

Page x of v



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Study Population: Safety Population

| Preferred Term | | | Test<br>Produc<br>N=XXX | t | | Comparator Placebo Product Product N=XXX N=XXX | | uct | Overall (N=XXX) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Intensity | n | (%) | [AEs] | n | (%) | [AEs] | n | (%) | [AEs] | n | (%) | [AEs] |
| Preferred Term #1 | MILD | XXX | (XX.X) | [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X) | [XXX] |
| | MODERATE | XXX | (XX.X) | [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X) | [XXX] |
| | SEVERE | XXX | (XX.X) | [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X) | [XXX] |
| Preferred Term #2 | MILD | xxx | (XX.X) | [XXX] | xxx | (XX.X | ) [XXX] | XXX | (XX.X | ) [XXX] | xxx | (XX.X) | [XXX] |
| | MODERATE | XXX | (XX.X) | [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X) | [XXX] |
| | SEVERE | XXX | (XX.X) | [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X | ) [XXX] | XXX | (XX.X) | [XXX] |
| Preferred Term #3 | MILD | xxx | (XX.X) | [777] | xxx | (VV V | ) [XXX] | VVV | (YY Y | ) [XXX] | vvv | (XX.X) | [VVV] |
| riciciled leim #5 | MODERATE | | | - | | | | | | | | | - |
| | | XXX | (XX.X) | - | XXX | | ) [XXX] | | | ) [XXX] | | (XX.X) | - |
| | SEVERE | XXX | (XX.X) | [XXX] | XXX | (AX.X | ) [XXX] | XXX | (AX.X | ) [XXX] | XXX | (XX.X) | [XXX] |

n (%) = Number (percent) of subjects nAE = Number of adverse events.

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD

Page x of v



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


 ${\tt Table~14.4.1.1}$  Summary of Oral Soft Tissue - Changes from Pre-treatment to Post-treatment Safety Population

Safety Population (N=xx)

| | | | | Post-Treatment (4 hours) | |
|---|---|---|---|---|---|
| | | | Normal | Abnormal | Not Examined |
| Treatment | AREA | Pre-Treatment | n (%) | n (%) | n (%) |
| Test Product | | | | | |
| | Labial Mucosa | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Not Examined | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Buccal Mucosa | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Not Examined | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | [other] | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | [oener] | Abnormal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Not Examined | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Comparator Product

Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD

Page x of v

Programmer Note: please add all different areas for all treatments.




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166

Listing 16.1.7.1

Randomization Details
All Randomized Subjects

Subject Number Age/Sex/ Race [1] Randomization Number Treatment Sequence [2] Randomization Date

Program Run Date:xxxx

Listing 16.1.7.1

Randomization Details
All Randomized Subjects

Randomization Date

PPD Page x of v

Programmer Note: correct seed number an block size to be added after unblinding in a footnote


<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

<sup>[2]</sup> A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.


| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.1.1 Subject Disposition All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| | | | | Treatment | Date of | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Age/Sex/ | Screening | Period | Start Date | Completion or | Period of | Completed | Primary Reason for | | |
| Number | Race [1] | Date | | and Time | Withdrawal | Withdrawal | (Yes/No) | Withdrawal | Further Details [2] | |
| | | | | | | | () | | | _ |

#### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

[2] Further details of reasons for withdrawal.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

#### PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

| B 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
|-----------------------------------------|----------------------|
| Protocol No. 208166 | Program Run Date:xxx |

Listing 16.2.1.2 Subject Disposition Non-Randomized Subjects

Subject
Number Age/Sex/ Race [1] Screening Date Reason for Screen Failure Further Details [2]

PPD

[2] Further details of reasons for screen failure.

PPD

<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166

Program Run Date:xxxx

Listing 16.2.2.1
Important and Major Protocol Deviations
All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject Number | Age/Sex/Race [1] | Period | Deviation Sequence | Date of Deviation | Deviation Type | Deviation Description |
|---|---|---|---|---|---|---|
| • | | | | | | _ |
| XXXXXX | XX/F/A1 | | 1 | 28JUN201 | XXXXXX | XXXXXX |

[1] Age in years; Sex: F=Female, M=Male; Race: A1=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD Page x of v

Programming Note: Listing 16.2.2.1 lists only those identified in population definition document to be excluded from PP population.



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Sodium fluoride and potassium nitrate 208166 Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.2.2

Minor Protocol Deviations
Randomized Population

xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx

Treatment Sequence: XXXXXXXXXX

Subject

Number Age/Sex/ Race [1] Period Deviation Sequence Protocol Deviation

PPD

African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

[1] Age in years; Sex: F=Female, M=Male; Race: A1=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.3.1
Exclusions from Analysis Populations
All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| | Age/Sex/ Race [1] | | | | |
|---|---|---|---|---|---|
| Subject Number | 1190,0011, 11000 [2] | Randomized | Safety | ITT | Per Protocol |

#### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.
A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

|-----------------------------|
| Listing 16.2.4.1 |
| Demographic Characteristics |
| All Randomized Subjects |

Treatment Sequence: XXXXXXXXXX

Subject Number

Race Age (years) Ethnicity

PPD

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.4.2 Medical History and Current Medical Conditions

All Randomized Subjects Treatment Sequence: XXXXXXXXXX

Subject Age/Sex/ Any Medical

Number Race [1] History? Medical Condition Start Date

PPD

Subject Age/Sex/ Any Medical Condition Start Date Ongoing? End Date

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD Page x of v



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.5.1

Prior Medications and Significant Non-Drug Therapies Prior to Treatment

All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject | Age/Sex/ Race [1] | Treatment | Reason for | Route of | Dose per | Frequency | Start Date | End Date/ |
|---|---|---|---|---|---|---|---|---|
| Number | | (GSK Drug | Medication | Administration | Administration | | (Study Day | Ongoing |
| | | Synonym) | | | | | [2]) | |

#### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

[2] Study day relative to the date of first dose of treatment.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.5.2

Concomitant Medications and Significant Non-Drug Therapies During Treatment

All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject<br>Number | Age/Sex/ Race [1] | Treatment<br>(GSK Drug | Medication assigned | Reason for<br>Medication | Route of<br>Administration | Dose per<br>Administration | Frequency | Start Date<br>(Study Day | End Date/<br>Ongoing |
|---|---|---|---|---|---|---|---|---|---|
| | | Synonym) | Period | | | | | [2]) | |

#### PPD

PPD Page x of y

Programmer Note: Subject will be listed by treatment groups. Same subjects could be listed on different treatment groups

GlaxoSmithKline Consumer Healthcare 

<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product

<sup>[2]</sup> Study day relative to the date of first dose of treatment.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Sodium fluoride and potassium nitrate 208166 Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166 Program Run Date:xxxx Listing 16.2.5.3 Study Product Compliance All Randomized Subjects Subject Number Age/Sex/ Race [1] Treatment Period Subject Compliance to use Number of missed Number of additional of washout period (Yes/No) product uses since the product uses since Sequence last visit the last visit

PPD

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD

<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.6.1 Surface Microhardness Recovery All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject | Age/Sex/ Race | Timepoint | Specimen | Period | Treatment | Measurement | Indentation | Indentation | Indentation | % SMHR |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | [1] | | Information | | | | length of | length after | length after in | |
| | | | | | | | sound enamel | first Erosive | situ | |
| | | | | | | | at baseline | Challenge | Remineralization | |
| | | | | | | | (B) | (E1) | (R) | |
| | | | | | | | ( u m) | ( u, m) | ( u m) | |

### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

Each value is calculated as the average of five indentations measurements per specimen, averaged across the four specimens for 2hours or 4hours.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD

Page x of y

Programmer Note: Please add all "other" information and timepoints for each subject in chronological order. For each subject we will have four specimen informations (XXXI to XXX4) per subject and period. Overall endpoint value to be calculated as mean of averages per period.

GlaxoSmithKline Consumer Healthcare 



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.6.2
Relative Erosion Resistance
All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

Subject Age/Sex/ Race Timepoint Specimen Period Treatment Measurement Sound First Erosive Indentation % RER Number [1] Information Enamel at Challenge length after Baseline second Erosive  $(\mu m)$ Challenge (E2) (μm) (μm)

### PPD

Each value is calculated as the average of five indentations measurements per specimen, averaged across the four specimens for 2hours or 4hours.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

#### PPD

Programmer Note: Please add all "other" information and timepoints for each subject in chronological order. For each subject we will have four specimen informations (XXXI to XXX4) per subject and period. Overall endpoint value to be calculated as mean of averages per period.


<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.6.3 Enamel Fluoride Uptake All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

Subject Age/Sex/ Race Timepoint Period Treatment Specimen Specimen Specimen Specimen Enamel Fluoride Number [1] Information Information Information Information Uptake

#### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: A1=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.6.4
Acid Resistance Ratio
All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject | Age/Sex/ | Timepoint | Specimen | Period | Treatment | Measurement | Sound | First | Second | In situ | Acid |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Race [1] | | Information | | | | Enamel at | Erosive | Erosive | Remineralization | Resistance |
| | | | | | | | Baseline | Challenge | Challenge | (μm) | Ratio |

#### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

Each value is calculated as the average of five indentations measurements per specimen, averaged across the four specimens for 2hours or 4hours.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

#### PPL

Page x of y

Programmer Note: Please add all "other" information and timepoints for each subject in chronological order. For each subject we will have four specimen informations (XXXI to XXX4) per subject and period. Overall endpoint value to be calculated as mean of averages per period.




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Organ Class]


Listing 16.2.7.1

Adverse Events

All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject<br>Number | Age/Sex/<br>Race [1] | Adverse Event (Preferred Term) [System of | Start Date<br>(Study<br>Day)[2] | Start<br>Time | End Date | End<br>Time | AE<br>assigned<br>Period | Frequency/ Intensity[3] | Related<br>to Study<br>Product? | Action<br>Taken re<br>Study<br>Product | Outcome | Seri<br>ous? | With-<br>drew?<br>[4] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

PPD

00 Adverse events with verbatim text ending in this are classified as Oral AEs.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD Page x of v

<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: A1=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

<sup>[2]</sup> Study day is the day relative to start of treatment, Day 1 being the day of first treatment. Period day is the day relative to the start of treatment being received in that period

<sup>[3]</sup> INT = Intermittent and SGLE = Single. [4] Did subject withdraw from study as a result of this adverse event?



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

Protocol No. 208166 Program Run Date:xxxx Listing 16.2.7.2

Adverse Events
Non-Randomized Subjects

Subject Age/Sex/ Adverse Event Start Date Start End Date End Frequency/ Related Action Outcome Seri With-Number Race [1] Time to Study Taken re drew? (Preferred Intensity[2] Product? Study [3] Term) Product [System of

[System of Organ Class]

PPD

@@ Adverse events with verbatim text ending in this are classified as Oral AEs.

PPD

<sup>[1]</sup> Age in years; Sex: F=Female, M=Male; Race: A1=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

<sup>[2]</sup> INT = Intermittent and SGLE = Single.

<sup>[3]</sup> Did subject withdraw from study as a result of this adverse event?



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.7.3 Listing of Incidents All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

Subject Number Age/Sex/Race[1] Treatment Period Date of the Incident Incident

#### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD



| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018

A=Test Product; B=Comparator Product; C=Placebo Product


Listing 16.2.9.1
Oral Soft Tissue Examination
All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject | Age/Sex/ Race [1] | Visit | Timepoint | Date of | Time of | Area | Abnormality | Details for not |
|---|---|---|---|---|---|---|---|---|
| Number | | | | Assessment | Assessment | | | examined |

## PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO3 plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD Page v of v




| Document Name | gsk-208166-reporting-and-analysis-plan-redact.pdf | |
|---|---|---|
| eldo controlled | 0.1; CURRENT; Most-Recent; In Review | 090032d58126e110 |
| Reason For Issue | | |

Statistical Reporting and Analysis Plan Amendment 1, 27 Feb 2018


Listing 16.2.9.2
Oral Hard Tissue Examination
All Randomized Subjects

Treatment Sequence: XXXXXXXXXX

| Subject | Age/Sex/ Race | Timepoint | Date of | Time of | Area | Abnormality | Details for not |
|---|---|---|---|---|---|---|---|
| Number | [1] | | Assessment | Assessment | | | examined |

### PPD

[1] Age in years; Sex: F=Female, M=Male; Race: Al=African American/African Heritage, A2=American Indian Or Alaskan Native, A3=Asian-Central/South Asian Heritage, A4=Asian-East Asian Heritage, A5=Asian-Japanese Heritage, A6=Asian-South East Asian Heritage, N=Native Hawaiian Or Other Pacific Islander, W1=White-Arabic/North African Heritage, W2=White-White/Caucasian/European Heritage, MT=Multiple.

A=Test Product; B=Comparator Product; C=Placebo Product

Test Product: Experimental dentifrice containing 0.254% w/w sodium fluoride (1 150 ppm fluoride) and 5% KNO<sub>3</sub> plus 0.25% PVM/MA copolymer and 2.5% sodium lactate; Comparator Product: Crest ProHealth Sensitivity & Enamel Shield dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride); Placebo Product: Fluoride free placebo dentifrice containing 5% KNO<sub>3</sub> (0 ppm fluoride); plus 0.25% PVM/MA copolymer and 2.5% lactate.

PPD